CLINICAL TRIAL: NCT03871231
Title: An International Clinical Feasibility Study to Evaluate the Safety and Performance of Low-Energy Unpinning Termination Therapy in Patients With VT/VF
Brief Title: Unpinning Termination Therapy for VT/VF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Cardialen, Inc. (Industry)
Collaborators: Genae (Industry); Five Corners (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL006
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
Keywords: Termination; Unpinning; Therapy
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: Non-randomized, non-blinded, prospective, single-arm, acute, early-feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Unpinning Termination Therapy Arm (Experimental): Subjects will have VT/VF induced and the Cardialen External Stimulation System (CESS) device will deliver electrical stimulation to terminate the arrhythmia
  Interventions: Device: Unpinning Termination Therapy

INTERVENTIONS:
Device: Unpinning Termination Therapy — The Cardialen External Stimulation System (CESS) is the research delivery system for the proprietary Cardialen Unpinning Therapy (UPT) therapy. The CESS is a custom designed and built research device. It is comprised of off-the-shelf commercial components (power supplies, waveform generators, laptop computer, monitor, rack, ECG system, leads, etc.) combined with a custom electrical circuit board and custom software.
  Other Names: Multi-pulse therapy; Multi-stage therapy; Multi-stage electrotherapy

SUMMARY:
This study is intended to develop a better method for stopping potentially lethal heart rhythms than currently available defibrillators. This new method, called Unpinning Termination Therapy (UPT), is hypothesized to be effective in stopping these dangerous heart rhythms at lower voltages and energy than current defibrillators. Consequently, UPT may improve survival, reduce patient pain from shocks, and lead to longer lasting and smaller implantable defibrillators.

DETAILED DESCRIPTION:
A prospective single-arm feasibility study involving acute testing of UPT electrotherapy in subjects with VT/VF during clinically indicated ventricular tachycardia catheter ablation procedure or indicated implantable cardioverter defibrillator implant, upgrade, or replacement or new CRT-D implant or upgrade to CRT-D.

The study involves up to two roll in subjects at each participating site followed by an UPT evaluation and refinement segment in which remaining subjects are enrolled until arrhythmia terminations from UPT delivery are reliably achieved. A prospective evaluation segment will be performed to compare UPT against SBS and ATP if sufficient subjects remain once reliable terminations from UPT are achieved.

Subjects will be evaluated at the visits for the Clinically-Indicated Procedure per standard of care. A single follow-up at up to 30 days post-procedure is required to assess subjects for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy of 1 year or greater
2. Male or female between 18 and 75 years of age
3. Willing and able to comply with the study protocol, provide a written informed consent
4. Indication for an endocardial VT catheter ablation for sustained, life-threatening monomorphic VT OR an indication for VF and ICD implant (de novo implant, replacement or upgrade) OR CRT-D (de novo implant, upgrade from ICD) with transvenous leads for the risk of or presence of VT and/or VF.
5. Etiology of arrhythmia, or risk of arrhythmia being ischemic dilated cardiomyopathy or non-ischemic idiopathic dilated cardiomyopathy both with LVEF ≤ 35% and meeting local standard of care
6. Medically stable at time of consent to undergo DFT testing performed under general anesthesia or conscious sedation as determined by the investigator

Exclusion Criteria:

The subject must not meet any of the following exclusion criteria:

1. Medically unstable at time of study and unsafe to undergo DFT testing under general anesthesia or conscious sedation as determined by the investigator
2. Hemodynamic instability as determined by the investigator
3. AF or atrial flutter for ≥ 48 hours or unknown duration, and no anticoagulation for preceding 3 weeks and no preoperative transesophageal echocardiographic confirmation of the absence of RA and LA thrombus
4. AF or atrial flutter for <48 hours and no Preoperative transesophageal echocardiographic confirmation of the absence of RA and LA thrombus
5. Presence of intracardiac thrombus
6. Inability to pass catheters to heart due to vascular limitations
7. Cardiovascular anatomical defects that would complicate placement of the lead or catheter required by the protocol, including congenital heart disease and cardiac vein anomalies as determined by the investigator
8. Pregnancy confirmed by test within 7 days of procedure
9. Pacemaker dependent
10. The presence of a normally functioning left ventricular lead which is not planned for revision
11. Presence of ventricular assist device, including Intra-aortic balloon pump
12. Subjects requiring the use of I.V. inotropes and/or vasopressors for hemodynamic support in the 14 days prior to the study
13. Prior VT catheter ablation with associated serious complication, such as hemodynamic compromise despite pressor agents, stroke, cardiac perforation, AC fistula, pneumothorax, sepsis
14. Incessant VT/VF or VT/VF storm
15. LVEF < 20%
16. New York Heart Association (NYHA) Class IV heart failure
17. Planned epicardial VT ablation on the same day as the research study
18. History of hyper-coagulable state that could increase risk of thromboembolic events
19. History of hemodynamic compromise due to valvular heart disease requiring IV inotropes or other circulatory support.
20. Unstable coronary artery disease as determined by the investigator
21. Severe proximal three-vessel or left main coronary artery disease, without revascularization as determined by the investigators
22. History of embolic stroke, Transient Ischemic Attack or other thromboembolic event in the past 6 months
23. History of Hypertrophic Cardiomyopathy, Arrhythmogenic Right Ventricular Dysplasia, Congenital Heart Anomaly, Cardiac Amyloidosis, Genetic Cardiac Channelopathy or Cardiac Sarcoidosis.
24. Cardiovascular surgery or intervention within 1 month prior to enrollment or planned for up to 1 month after enrollment (other than the planned treatment procedure)
25. Morbid obesity: BMI>39 kg/m2
26. Cognitive or mental health status that would interfere with study participation and proper informed consent
27. Presence of mechanical tricuspid valve
28. Active Endocarditis
29. Ventricular arrhythmia etiology sarcoidosis
30. Valvular ventricular tachycardia
31. Previously implanted lead is under recall by manufacturer or evidence of lead failure as determined by the investigator
32. End Stage Renal Disease on hemodialysis or peritoneal dialysis, or estimated glomerular filtration rate (eGFR) <15 ml/min
33. Right atrial or right ventricular lead implanted within 12 months prior to screening
34. Any other medical condition which may affect the outcome of this study or safety of the subject as determined by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Safety of UPT therapy | Study procedure and 30 day post procedure
  Adverse events
Safety of UPT therapy | 30 day post procedure
  Adverse events
Parameters at which UPT terminates VT and VF | Study procedure
  Voltage

SECONDARY OUTCOMES:
Voltage at which UPT and endocardial single biphasic shock terminate VT/VF | Study procedure
  Voltage
Voltage at which UPT and ATP terminate VT | Study procedure
  Voltage

CONTACTS AND LOCATIONS:
Overall Officials: Harris Haqqani, MD, Principal Investigator — The Prince Charles Hospital
Locations (4):
- Australia (4):
  - The Prince Charles Hospital, Chermside, Queensland
  - Gold Coast, Southport, Queensland
  - Royal Adelaide Hospital, Norwood, South Australia
  - Monash Medical, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janardhan AH, Gutbrod SR, Li W, Lang D, Schuessler RB, Efimov IR. Multistage electrotherapy delivered through chronically-implanted leads terminates atrial fibrillation with lower energy than a single biphasic shock. J Am Coll Cardiol. 2014 Jan 7-14;63(1):40-8. doi: 10.1016/j.jacc.2013.07.098. Epub 2013 Sep 26. PMID 24076284
- [Background] Janardhan AH, Li W, Fedorov VV, Yeung M, Wallendorf MJ, Schuessler RB, Efimov IR. A novel low-energy electrotherapy that terminates ventricular tachycardia with lower energy than a biphasic shock when antitachycardia pacing fails. J Am Coll Cardiol. 2012 Dec 11;60(23):2393-8. doi: 10.1016/j.jacc.2012.08.1001. Epub 2012 Nov 7. PMID 23141483
- [Background] Li W, Janardhan AH, Fedorov VV, Sha Q, Schuessler RB, Efimov IR. Low-energy multistage atrial defibrillation therapy terminates atrial fibrillation with less energy than a single shock. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):917-25. doi: 10.1161/CIRCEP.111.965830. Epub 2011 Oct 6. PMID 21980076
- [Background] Efimov I, Ripplinger CM. Virtual electrode hypothesis of defibrillation. Heart Rhythm. 2006 Sep;3(9):1100-2. doi: 10.1016/j.hrthm.2006.03.005. Epub 2006 Mar 10. No abstract available. PMID 16945810
- [Background] Ripplinger CM, Krinsky VI, Nikolski VP, Efimov IR. Mechanisms of unpinning and termination of ventricular tachycardia. Am J Physiol Heart Circ Physiol. 2006 Jul;291(1):H184-92. doi: 10.1152/ajpheart.01300.2005. Epub 2006 Feb 24. PMID 16501014
- [Background] Li W, Ripplinger CM, Lou Q, Efimov IR. Multiple monophasic shocks improve electrotherapy of ventricular tachycardia in a rabbit model of chronic infarction. Heart Rhythm. 2009 Jul;6(7):1020-7. doi: 10.1016/j.hrthm.2009.03.015. Epub 2009 Mar 11. PMID 19560090
- [Background] Ambrosi CM, Ripplinger CM, Efimov IR, Fedorov VV. Termination of sustained atrial flutter and fibrillation using low-voltage multiple-shock therapy. Heart Rhythm. 2011 Jan;8(1):101-8. doi: 10.1016/j.hrthm.2010.10.018. Epub 2010 Oct 19. PMID 20969974